CLINICAL TRIAL: NCT01700465
Title: Estimating and Predicting Hemodynamic Changes During Hemodialysis
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 11-1437
Record Dates: First submitted 2012-09-27; First posted 2012-10-04 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Hemodialysis
Keywords: Hemodialysis; Hemodynamics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hemodialysis: Patients undergoing hemodialysis

SUMMARY:
Machine learning techniques and algorithms originally developed for use in the field of robotics can be applied to continuous, noninvasive physiological waveform data to discover hidden, hemodynamic relationships. Newly developed algorithms can, in real-time: 1) estimate acute blood loss volume, 2) monitor and estimate fluid resuscitation needs, 3) predict cardiovascular collapse well ahead of any clinically significant changes in standard vital signs, and 4) estimate intracranial pressure. We hypothesize that these same methods can be used to monitor volume loss during hemodialysis, as well as predict intradialytic hypotension, well before it occurs.

DETAILED DESCRIPTION:
1. Collect physiological waveform data from patients undergoing hemodialysis at the University of Colorado Hospital, Children's Hospital Colorado, and Fresenius Medical Centers using non-invasive monitoring techniques.
2. Combine the physiological data from patient monitors with clinical and demographic data, including age, gender, race, problem list, reason for dialysis, estimated dry weight, volume removed, arterial and venous pressures, etc. for use in developing mathematical models of hemodialysis.
3. Develop robust, real-time, computational models for:

   * estimating acute intravascular volume loss during hemodialysis
   * predicting an optimal, individual specific, intravascular volume to be removed during a hemodialysis session
   * predicting intradialytic hypotension
4. Determine:

   * which non-invasive signals are relevant to each model type
   * which features extracted from these signals are relevant
   * which algorithms are capable of using the extracted features for each decision type

ELIGIBILITY:
Inclusion Criteria:

* Age: 2 - 89 years
* Undergoing hemodialysis at the Fresenius Medical Centers, University of Colorado Hospital or Children's Hospital Colorado

Exclusion Criteria:

* Pregnant
* Incarcerated
* Decisionally challenged
* Positive for hepatitis B surface antigen
* Limited access to or compromised monitoring sites for non-invasive finger and ear or forehead sensors

Ages: 2 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult and pediatric patients undergoing hemodialysis at Fresenius Medical Centers, University of Colorado Hospital or Children's Hospital Colorado will be the population base for enrollment in this study. Patients may have acute kidney injury or end stage renal disease. Subjects may be inpatients or outpatients.
Sampling Method: Non-Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2012-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Acute intravascular volume loss during hemodialysis | one hemodialysis session (approx 3-4 hours)
  development of algorithm to estimate acute intravascular volume loss during hemodialysis

CONTACTS AND LOCATIONS:
Overall Officials: Steve Moulton, MD, Principal Investigator — Children's Hospital Colorado
Locations (5):
- United States (5):
  - Fresenius Medical Center East Denver, Aurora, Colorado
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Fresenius Medical Center Central, Denver, Colorado
  - Fresenius Medical Center Rocky Mountain, Denver, Colorado